CLINICAL TRIAL: NCT06253702
Title: Human Cerebral Blood Flow Regulation: Sex, Mechanism, and Stress Differences (Phase 2)
Brief Title: Brain Blood Flow Responses to Stress: Sex Differences
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023-0548; 1R01HL150361-01 (NIH); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 07/01/2024 (Other: UW Madison)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cerebrovascular Disorders
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Indomethacin; elagolix; Anastrozole; Estradiol

STUDY DESIGN:
Intervention Model Description: double-blind placebo controlled design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo First: Hormone Suppression (Experimental): Participants drug (placebo vs Indo) are randomized prior to first set of MRI visits, while experiencing hormone suppression.
  Interventions: Drug: Indomethacin; Drug: Placebo; Drug: Orilissa; Drug: Estradiol
- Indo First: Hormone Suppression (Experimental): Participants drug (placebo vs Indo) are randomized prior to first set of MRI visits, while experiencing hormone suppression.
  Interventions: Drug: Indomethacin; Drug: Placebo; Drug: Orilissa
- Placebo First: Hormone Add-Back (Experimental): Participants drug (placebo vs Indo) are randomized prior to second set of MRI visits, while experiencing hormone add-back.
  Interventions: Drug: Indomethacin; Drug: Placebo; Drug: Orilissa; Drug: Testosterone gel; Drug: Anastrozole; Drug: Estradiol
- Indo First: Hormone Add-Back (Experimental): Participants drug (placebo vs Indo) are randomized prior to second set of MRI visits, while experiencing hormone add-back.
  Interventions: Drug: Indomethacin; Drug: Placebo; Drug: Orilissa; Drug: Testosterone gel; Drug: Anastrozole; Drug: Estradiol

INTERVENTIONS:
Drug: Indomethacin — to inhibit cyclooxygenase (COX)
  Other Names: Indo
Drug: Placebo — Placebo
Drug: Orilissa — to suppress hormones 200mg dose 2x per day (all participants)
Drug: Testosterone gel — 50 mg each morning for add back phase (male participants)
  Arms: Indo First: Hormone Add-Back; Placebo First: Hormone Add-Back
Drug: Anastrozole — 1mg/day in men to prevent conversion of testosterone to estradiol
  Arms: Indo First: Hormone Add-Back; Placebo First: Hormone Add-Back
Drug: Estradiol — Women will receive oral estradiol 2mg/daily
  Arms: Indo First: Hormone Add-Back; Placebo First: Hormone Add-Back; Placebo First: Hormone Suppression

SUMMARY:
Twenty-six otherwise healthy adults between 18-40 years of age composed of 13 males and 13 females will be enrolled in this study to determine how sex and sex hormones influence cerebral blood flow (CBF) control in healthy young adults without confounds of age or disease. Participants can expect to be on study for approximately 16 days.

DETAILED DESCRIPTION:
Objective: To determine cerebrovascular control mechanisms in humans and provide mechanistic knowledge to offer new sex-specific therapeutic options for cerebrovascular diseases. The current objective is to determine how sex and sex hormones influence CBF control in healthy young adults without confounds of age or disease.

The central hypothesis is men exhibit reduced cerebral vasodilator function due in part to differences in COX signaling compared to women. Comprehensive CBF data from multi-modal MRI indicate the magnitude of sex differences-as well as the vasodilator mechanisms-are regionally distinct.

The investigators will address 2 specific aims:

1. Are cerebral vasodilator responses greater in women across other physiologic stressors? Do all cerebral vessels respond equally, or are there regional differences-by sex?
2. What mechanisms regulate the increase in CBF to stress; do these differ by sex, or brain region?

This study will be conducted in compliance with federal investigational drug regulations (21 CFR 312) and Good Clinical Practice (GCP) guidelines, as well as state law and institutional policies.

Study Population: Phase 2 include 26 total participants 13 men and 13 women invited back from the Study 2020-0336 (NCT04265053) for Aim 3 who are ≥18 - ≤ 40 years old and considered healthy.

Approach: CBF testing will be performed in research-dedicated 3T magnets. Participants will experience one hypoxia and one hypercapnia trial during each visit. S, study design focuses on the use of Indomethacin to test COX as a potential mechanism explaining sex differences in CBF control. To do this, 4 MRI visits in a double-blind placebo controlled design will be conducted. One set of placebo-Indo visits occurs after the first 4-7 days of sex hormone suppression (with Orilissa) and the second set of MRI visits occurs after 12-16 days of Orilissa while supplementing a single sex hormone by sex.

On day 0 participants will start hormone suppression using Orilissa (male subjects will also start an Anastrozole). After day 2, MRI Visit 1 will be scheduled to occur. Prior to the first study visit the order of drug supplementation will be randomized. Options are: placebo for the first MRI visit, then Indomethacin for the second MRI visit or Indomethacin for the first MRI visit, then placebo for the second MRI visit. After MRI visits 1 and 2 are completed, participants will begin sex hormone add-back (males will receive testosterone and females will receive estradiol). Once participants have been on the hormone add-back protocol for 3-4 days MRI Visits 3 and 4 will be scheduled. Prior to MRI visit 3 the order of drug supplementation will be randomized again.

. Added to protocol on 07/01/2024 = Fecal samples will be collected: at baseline (before beginning Orilissa), 4-8 days after taking the first dose of Orilissa, and 12-16 days after taking the first estradiol or testosterone dose. Subjects will provide 3 fecal samples at home throughout the course of their participation and will take the samples to FedEx to be shipped.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥18 - ≤40 years inclusive
* Completed Phase 1: Study 2020-0336

Exclusion Criteria:

* Hypertensive

  * > 125 mmHg systolic blood pressure; or
  * > 80 mmHg diastolic blood pressure
* BMI ≥25 kg/m2
* Fasting blood glucose ≥100 mg/dl
* LDL cholesterol ≥130 mg/dl
* Triglycerides ≥150 mg/dl
* Current diagnosis or history of:

  * peripheral vascular disease
  * hepatic disease
  * renal disease
  * lung disease
  * gastrointestinal disorders/bleeding
  * hematologic disease
  * stroke
  * myocardial infarction
  * coronary heart disease
  * congestive heart failure
  * heart surgery
  * prediabetes
  * diabetes mellitus (type 1, type 2, MODY, or others)
  * sleep apnea
  * hypertension
  * some autoimmune diseases, such as inflammatory bowel disease or systemic lupus erythematosus (exclusion at discretion of reviewing MD)
* Current smoking, defined as the use of tobacco or nicotine products >5 times in the past 30 days.
* Cardiovascular medication use
* NSAID sensitivity
* Magnesium-restricted diet
* Any contraindications of having an MRI

  * (e.g. the requirement of anxiolytics in order to complete an MRI scan)
* Irregular menstrual cycle (females only)
* Medical conditions that can affect the menstrual cycle, such as hyperprolactinemia, prolactinoma, hypercortisolemia, and congenital adrenal hyperplasia (females only)
* Pregnancy, breast feeding, or plans to conceive within the next 3 months (females only)
* Polycystic ovary syndrome (females only)
* Hirsutism defined as unwanted and/or excessive hair growth on the face, chest, or back (females only)
* Levonorgestrel intrauterine device (IUD) (females only)
* Hormonal birth control will not be allowed in women, in order to control for high variability between type, dose, and route of therapy. However, in discussion with Dr. Davis (Co-I) and Dr. Laura Cooney M.D., physician experts in medical and reproductive endocrinology and infertility, there are two broad exceptions to this birth control criteria:

  * Copper intrauterine devices (IUDs) will be allowed as they do not change systemic sex hormone levels).
  * Women currently taking hormonal birth control (i.e. contraceptive pills, patch, ring) for contraception only (not for a medical condition such as those listed in exclusion criteria above) may consider temporarily stopping to become eligible for enrollment. Hormonal birth control must be stopped at least one month prior to Study Visit 1 to provide time for menstruation to resume. Then stoppage continues through the last planned study visit. Screening information will be reviewed by endocrinology physicians to determine eligibility and timing on this issue.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Cerebral Blow Flow (CBF): Hormone Suppression Hypoxia Condition | first set of study visits (up to 2 hours) within the first 7 days on study
  Hypoxia condition will be measured twice via MRI during the first set of study visits under hormone suppression. Reported here is the CBF under hypoxia for the placebo group as compared to the CBF under hypoxia for the Indo group.
Cerebral Blow Flow: Hormone Suppression Hypercapnia Condition | first set of study visits (up to 2 hours) within the first 7 days on study
  Hypercapnia condition will be measured twice via MRI during the first set of study visits under hormone suppression. Reported here is the CBF under hypercapnia for the placebo group as compared to the CBF under hypercapnia for the Indo group.
Cerebral Blow Flow: Hormone Add-Back Hypoxia Condition | second set of study visits (up to 2 hours) within 12-16 days on study
  Hypoxia condition will be measured twice via MRI during the second set of study visits under hormone add-back. Reported here is the CBF under hypoxia for the placebo group as compared to the CBF under hypoxia for the Indo group.
Cerebral Blow Flow: Hormone Add-Back Hypercapnia Condition | second set of study visits (up to 2 hours) within 12-16 days on study
  Hypercapnia condition will be measured twice via MRI during the first set of study visits under hormone add-back. Reported here is the CBF under hypercapnia for the placebo group as compared to the CBF under hypercapnia for the Indo group.

CONTACTS AND LOCATIONS:
Overall Officials: William G Schrage, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No